CLINICAL TRIAL: NCT04238221
Title: Effect of Doxofylline on Bronchial Obstruction, in add-on to Maximal Inhalation Therapy, in Clinically Stable COPD Patients.
Brief Title: Effect of add-on Doxofylline on Lung Function in Stable COPD
Acronym: EDAI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Pierachille Santus, MD, PhD, Professor of Respiratory Diseases, Head of the Respiratory Disease Unit, L. Sacco University Hospital, Milan, Italy, University of Milan
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 01-PNSNP-2020
Record Dates: First submitted 2020-01-14; First posted 2020-01-23 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Bronchodilator; Pulmonary Function Test; Doxofylline; Methylxanthines; 6-minute walk test; FEV1
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — doxofylline

STUDY DESIGN:
Intervention Model Description: Phase 4, single center, prospective, interventional, randomized, single blind, crossover
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization, drug administration and patient training will be performed by an operator not involved in patients' recruitment and in the data collection and analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Doxofylline+inhalation therapy (Experimental): 4-week treatment with doxofylline tablets 400 mg bid in addition to maximal inhalation therapy, followed by 4-week treatment of maximal inhalation therapy only
  Interventions: Drug: Doxofylline
- Inhalation therapy (Experimental): 4-week treatment with maximal inhalation therapy only, followed by 4-week treatment with doxofylline tablets 400 mg bid in addition to maximal inhalation therapy
  Interventions: Drug: Doxofylline

INTERVENTIONS:
Drug: Doxofylline — Patients will receive a 4-week treatment with doxofylline 400 mg bid, in addition to their chronic usual inhalation therapy.
  Other Names: Ansimar

SUMMARY:
It is a phase IV, prospective, interventional, single blind, randomized, crossover trial in which the investigators will evaluate the effects of a 4-week treatment with doxofylline 400 mg bid, in add-on to maximal inhalation therapy, in clinically stable COPD patients.

DETAILED DESCRIPTION:
The investigators will evaluate the effects of a 4-week treatment with doxofylline 400 mg, in add-on to maximal inhalation therapy (bronchodilators with or without a fixed dose combination with inhaled corticosteroids), in clinically stable COPD patients.

After screening and collection of informed consent, study participants will undergo a 7-day run-in, during which compliance to inhaled therapy and clinical stability will be assessed.

On the first visit patients will complete questionnaires (CAT, mMRC and SGRQ) to assess baseline respiratory function and health related quality of life.

After the first visit, patients will undergo a washout period during which the inhaled therapy will be withheld for 24 hours (7 days in case of chronic therapy with tiotropium).

The following day (the 8th day in case of tiotropium use), patients will perform the baseline measurement of the following:

1. plethysmography
2. DLCO
3. maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP)
4. 6-minute walk test (6MWT) with the assessment of dyspnea scale (Borg scale) at rest and after exercise.

Sixty minutes after the administration of the usual chronic inhalation therapy, patients will then perform the same respiratory lung functional bundle of tests as detailed above (from 1 to 3).

Subsequently, patients will be randomized in two parallel arms (arm A and arm B). Patients assigned to arm A will be prescribed 30-day treatment with doxofylline 400 mg bid, in addition to their chronic inhalation therapy, and will take the first dose of the medication; patients assigned to arm B will have their chronic therapy unchanged.

Randomization, drug administration and patient training will be performed by an operator not involved in patients' recruitment, data collection and analysis.

180 minutes after the administration of the usual chronic inhalation therapy, patients will repeat the lung function bundle from point 1 to 3.

During the subsequent 4-week treatment, patients' compliance will be monitored by telephone calls. Any adverse event will be registered and will be treated according to our center's standard operating procedures and good clinical practice by the treating physician.

After 4 weeks, before the administration of the morning dose, patients will be asked to complete the CAT, mMRC and SGRQ questionnaires and to perform the baseline functional bundle detailed in points 1 to 4. Patients will be asked to take the home inhalation therapy, as well as doxofylline if arm A. Respiratory function tests from points 1 to 3 will be repeated 60 minutes after drug administration. After that, patients assigned to Arm B will take the first dose of doxofylline. Respiratory function tests from points 1 to 3 will then be repeated 180 minutes after inhalation therapy administration. Eventually, the 6-MWT will be performed by patients assigned to Arm A, with assessment of the Borg dyspnea scale.

During the subsequent 4 weeks, patients assigned to arm B will be prescribed therapy with doxofylline 400 mg bid in addition to their chronic inhalatory therapy, while patients assigned to arm A will have only their usual chronic inhalation therapy. Compliance monitoring and adverse event management will be handled as previously discussed.

At the end of the 4 weeks, before the administration of the morning dose, patients will be asked to complete the CAT, mMRC and SGRQ questionnaires and to perform the baseline functional bundle detailed in points 1 to 4. Patients will be asked to take the home inhalation therapy, as well as doxofylline if arm B. Respiratory function tests from points 1 to 3 will be repeated 60 minutes and 180 minutes after drug administration. Eventually, the 6-MWT will be performed by patients assigned to Arm B, with assessment of the Borg dyspnea scale.

A 30-day follow up will be performed after the last visit, in order to register any late drug adverse reaction or adverse events..

ELIGIBILITY:
Inclusion Criteria:

* COPD diagnosis for at least 6 months, according to current European Respiratory Society guidelines
* baseline FEV1 ≤ 80% of predicted value
* active or former smokers with smoking history ≥ 10 pack-years
* patients chronically treated with a long acting muscarinic antagonist (LAMA) and a long acting beta-2 agonists (LABA), in association with or without an inhaled corticosteroid (ICS)
* clinically stable disease for 6 months.

Exclusion Criteria:

* previous or current diagnosis of bronchial asthma
* previous lung volume reduction through surgery or endobronchial valves
* inability to perform respiratory function tests according to international standards, or contraindications to perform 6-minute walking test
* known allergy or intolerance to doxofylline
* current or potential pregnancy
* mini-Mental test <21
* congestive heart failure NYHA III or IV
* recent (<6 months) myocardial infarction
* unstable arrhythmias
* chronic hypotension
* active peptic ulcer
* severe liver disease
* active neoplasia
* history of drug or alcohol abuse.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2020-10-30 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
Difference in changes in FEV1 after 4 weeks of treatment | 4-8 weeks
  Difference between changes in the Forced Expiratory Volume in one second (FEV1) measured at baseline and the FEV1 after 4 weeks of treatment with doxofylline in addition to inhalation therapy, measured 30 minutes before the morning dose of doxofylline plus inhalation therapy, and changes in the FEV1 measured at baseline and the FEV1 after 4 weeks of treatment with inhalation therapy only, measured 30 minutes before the morning dose of inhalation therapy.

SECONDARY OUTCOMES:
Change in FEV1 60' after drug administration | 60 minutes
  Changes in the Forced Expiratory Volume in one second (FEV1) measured at baseline and the FEV1 measured 60 minutes after the first dose of doxofylline plus inhalation therapy.
Difference in changes in distance covered in 6-minute walking test after 4 weeks of treatment | 4-8 weeks
  Difference between changes in the distance covered in the 6-minute walking test (6-MWT) performed at baseline and the distance covered in 6-MWT performed after 4 weeks of treatment with doxofylline in addition to inhalation therapy, 30 minutes before the morning dose of doxofylline plus inhalation therapy, and changes in the distance covered in the 6-MWT performed at baseline and the 6-MWT performed after 4 weeks of treatment with inhalation therapy alone, 30 minutes before the morning dose of inhalation therapy.
Changes in distance covered in 6-minute walking test 180' after drug administration | 4-8 weeks
  Change in the distance covered in the 6-minute walking test (6-MWT) performed at baseline and the distance covered in 6-MWT performed after 4 weeks of treatment with doxofylline in addition to inhalation therapy, 180 minutes after the morning dose of doxofylline
Difference in changes in resting and effort dyspnea after 4 weeks of treatment | 4-8 weeks
  Difference between changes in the modified Borg dyspnea scale assessed before and after the 6-minute walking test (6-MWT) performed at baseline and the modified Borg dyspnea scale assessed before and after the 6-MWT performed after 4 weeks of treatment with doxofylline in addition to inhalation therapy, 30 minutes before the morning dose of doxofylline plus inhalation therapy, and changes in the modified Borg dyspnea scale assessed before and after the 6-MWT performed at baseline and the modified Borg dyspnea scale assessed before and after the 6-MWT performed after 4 weeks of treatment with inhalation therapy alone, 30 minutes before the morning dose of inhalation therapy.
  Modified Borg dyspnea scale is used to rate difficulty of breathing and ranges from 0 (absence of dyspnea) to 10 (maximum dyspnea).
Changes in resting and effort dyspnea 180' after drug administration | 4-8 weeks
  Difference between the modified Borg dyspnea scale assessed before and after the 6-minute walking test (6-MWT) performed at baseline and the modified Borg dyspnea scale assessed before and after the 6-MWT performed after 4 weeks of treatment with doxofylline in addition to inhalation therapy, 180 minutes after the morning dose of doxofylline plus inhalation therapy.
  Modified Borg dyspnea scale is used to rate difficulty of breathing and ranges from 0 (absence of dyspnea) to 10 (maximum dyspnea).
Difference in changes in modified Medical Research Council (mMRC) scale after 4 weeks of treatment | 4-8 weeks
  Difference between changes in the score of modified Medical Research Council (mMRC) scale at baseline and after 4 weeks of treatment with doxofylline in addition to chronic inhalation therapy and changes in the score of mMRC at baseline and after 4 weeks of treatment with chronic inhalation therapy alone.
  The mMRC scale is used to assess the severity of dyspnea and ranges from 0 to 4; the higher the score, the higher the dyspnea sensation.
Difference in changes in COPD Assessment Test (CAT) score after 4 weeks of treatment | 4-8 weeks
  Difference between changes in the score of COPD Assessment Test (CAT) at baseline and after 4 weeks of treatment with doxofylline in addition to chronic inhalation therapy and changes in the score of CAT at baseline and after 4 weeks of treatment with chronic inhalation therapy alone.
  The CAT score is used to assess the impact of COPD on a patient's daily life, and ranges from 0 (suggesting no significant impact) to 40 (suggesting a very severe impact)
Difference in changes in St. George Respiratory Questionnaire (SGRQ) after 4 weeks of treatment | 4-8 weeks
  Difference between changes in the score of St. George Respiratory Questionnaire (SGRQ) at baseline and the score of SGRQ after 4 weeks of treatment with doxofylline in addition to inhalation therapy and changes in the score of SGRQ at baseline and the SGRQ after 4 weeks of treatment with inhalation therapy alone.
  SGRQ is designed to measure the impact on overall health, daily life, and perceived well-being in patients with obstructive airways disease. Scores range from 0 to 100, with higher scores indicating more limitations.
Difference in changes in vital capacity after 4 weeks of treatment | 4-8 weeks
  Difference between changes in the slow vital capacity (VC) measured at baseline and the VC after 4 weeks of treatment with doxofylline in addition to inhalation therapy, measured 30 minutes before the morning dose of doxofylline plus inhalation therapy, and changes in the VC measured at baseline and the VC after 4 weeks of treatment with inhalation therapy only, measured 30 minutes before the morning dose of inhalation therapy.
Difference in changes in residual volume after 4 weeks of treatment | 4-8 weeks
  Difference between changes in the residual volume (RV) measured at baseline and the RV after 4 weeks of treatment with doxofylline in addition to inhalation therapy, measured 30 minutes before the morning dose of doxofylline plus inhalation therapy, and changes in the RV measured at baseline and the RV after 4 weeks of treatment with inhalation therapy only, measured 30 minutes before the morning dose of inhalation therapy.
Difference in changes in functional residual capacity after 4 weeks of treatment | 4-8 weeks
  Difference between changes in the functional residual capacity (FRC) measured at baseline and the FRC after 4 weeks of treatment with doxofylline in addition to inhalation therapy, measured 30 minutes before the morning dose of doxofylline plus inhalation therapy, and changes in the FRC measured at baseline and the FRC after 4 weeks of treatment with inhalation therapy only, measured 30 minutes before the morning dose of inhalation therapy.
Difference in changes in inspiratory capacity after 4 weeks of treatment | 4-8 weeks
  Difference between changes in the inspiratory capacity (IC) measured at baseline and the IC after 4 weeks of treatment with doxofylline in addition to inhalation therapy, measured 30 minutes before the morning dose of doxofylline plus inhalation therapy, and changes in the IC measured at baseline and the IC after 4 weeks of treatment with inhalation therapy only, measured 30 minutes before the morning dose of inhalation therapy.
Difference in changes in specific airway resistance after 4 weeks of treatment | 4-8 weeks
  Difference between changes in the specific airway resistances (sRaw) measured at baseline and the sRaw after 4 weeks of treatment with doxofylline in addition to inhalation therapy, measured 30 minutes before the morning dose of doxofylline plus inhalation therapy, and changes in the sRaw measured at baseline and the sRaw after 4 weeks of treatment with inhalation therapy only, measured 30 minutes before the morning dose of inhalation therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- L. Sacco Hospital, Milan, Italy

IPD SHARING:
Plan to Share IPD: No